CLINICAL TRIAL: NCT00522756
Title: Preventing Acute Renal Failure After Cardiac Surgery in High Risk Patients Using Sodium Bicarbonate Therapy (PARACHUTE) - Pilot Study
Brief Title: Preventing Acute Renal Failure After Cardiac Surgery in High Risk Patients Using Sodium Bicarbonate Therapy
Acronym: PARACHUTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SDR-05-045
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Failure, Acute
Keywords: Kidney Failure, Acute; Cardiac Surgical Procedures; Sodium Bicarbonate; Sodium Chloride; Prevention and control
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Three ampoules of 7.5% sodium bicarbonate (89.3 mOsm/ampoule; total 150 ml for three ampoules) added to 750 ml of 5% dextrose in water, given at 1 ml/kg/hour through a dedicated intravenous line for 6 hours, and completed prior to the initiation of cardiopulmonary bypass.
  Interventions: Drug: Sodium bicarbonate
- Control (Active Comparator): 0.9% sodium chloride given at 1 ml/kg/hour through a dedicated intravenous line for 6 hours, and completed prior to the initiation of cardiopulmonary bypass.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium bicarbonate — Three ampoules of 7.5% sodium bicarbonate (89.3 mOsm/ampoule; total 150 ml for three ampoules) added to 750 ml of 5% dextrose in water, given at 1 ml/kg/hour through a dedicated intravenous line for 6 hours, and completed prior to the initiation of cardiopulmonary bypass.
  Other Names: NaHCO3
  Arms: Intervention
Drug: Sodium chloride — 0.9% sodium chloride given at 1 ml/kg/hour through a dedicated intravenous line for 6 hours, and completed prior to the initiation of cardiopulmonary bypass.
  Other Names: saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether sodium bicarbonate is effective in reducing kidney injury that may occur during cardiac surgery.

DETAILED DESCRIPTION:
Acute renal failure (ARF) is an important complication after cardiac surgery that has a prevalence ranging between 5 and 30%. In addition, the impact of chronic kidney disease (CKD) has been well correlated with poorer outcomes after cardiac surgery. These factors have been demonstrated to be associated with increased morbidity, mortality, as well as consuming limited health care resources.

Despite the identification of certain higher risk determinants such as emergency surgery, valvular surgery, preoperative creatinine level, diabetes, increasing age, obesity, and peripheral vascular disease, interventions to decrease postoperative ARF in these patients have been limited. Agents that have been successful in other settings, such as N-acetylcysteine and fenoldopam, have shown no difference in clinical outcomes of ARF when tested in randomized clinical trials in high-risk cardiac surgery patients. Although prophylactic hemodialysis has been shown to be effective for patients with underlying severe kidney disease, this is clearly a resource intensive therapy that may not be practical as a general prophylaxis strategy.

The use of sodium bicarbonate has shown efficacy in reducing the incidence of ARF due to contrast-induced nephropathy in those patients with moderate, stable renal dysfunction. The postulated mechanism of renal protection has been described through the prevention of free radical generation and damage. The generation of a higher renal proximal tubule pH with bicarbonate therapy may slow down the superoxide-generating Haber-Weiss reaction, limiting the formation of free radical oxidants. In addition, sodium bicarbonate may be directly scavenging reactive oxygen species generated from nitric oxide, at a physiologic pH.

If it is presumed that initiation and extension of ischemic renal injury occurs during cardiac surgery via oxidant injury, the use of sodium bicarbonate to disrupt this process could possibly be an effective therapeutic option to prevent ARF.

The objective of this study is to evaluate the renal protective effect of near-isotonic sodium bicarbonate as compared to sodium chloride when given as prophylaxis to patients with chronic kidney disease prior to non-emergent surgery involving the use of cardiopulmonary bypass.

Our hypothesis is that bicarbonate therapy may disrupt ischemia-induced, oxidant-mediated injury and this may prevent the propagation of renal damage. These events may be demonstrated clinically by a reduced incidence of ARF following surgery, decreased requirements for renal replacement therapy after surgery, and improved survival both perioperatively and in a longer-term follow up.

ELIGIBILITY:
Inclusion criteria:

* age greater than or equal to 18 years
* elective or urgent CABG +/- valve surgery, or elective or urgent isolated valve surgery
* exposure to cardiopulmonary bypass
* stable kidney disease: less than 25% change in serum creatinine during 3 months before surgery
* Estimated glomerular filtration rate, by Modification of Diet in Renal Disease (MDRD) equation, less than or equal to 60 ml/min/1.73m2

Exclusion criteria:

* emergency CABG, cardiac transplantation, or insertion of VAD
* planned off-pump surgery
* N-acetylcysteine given in last 72 hours prior to operation
* radiocontrast given in last 48 hours prior to operation
* acute renal failure (greater than 25% increase in serum creatinine from preadmission baseline)
* glomerular filtration rate less than 15 ml/min or chronic dialysis
* prior renal transplantation
* enrollment in another research study, with the exception of MUHC study SDR-05-033
* LV ejection fraction less than or equal to 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Increase in serum creatinine of 44 micromol/L or by 25% within the first 3 days after surgery. | 3 days

SECONDARY OUTCOMES:
Postoperative vasoactive medication, intra-aortic balloon pump, mechanical ventilation, reintubation, reoperation, myocardial infarction, stroke, infection, hypokalemia, dialysis, ICU and hospital length of stay and survival. | 3 weeks post operative period

CONTACTS AND LOCATIONS:
Overall Officials: Benoit de Varennes, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Ahsan Alam, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204